CLINICAL TRIAL: NCT06513858
Title: Evaluating the Impact of Community-Based Mindfulness and Musical Programs on Psychiatric Measures, Drum Circle Study 2c.
Brief Title: Evaluating the Community Drum Circle
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000028866_c; 2R25MH071584-11 (NIH)
Record Dates: First submitted 2024-07-10; First posted 2024-07-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Mental Health Issue; COVID-19
Keywords: Mindfulness; Meditation; Music
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drum Circle- Cohort 1 (Experimental): Cohort 1 will listen together to recordings of drumming and be allowed to drum along while listening.
  The facilitator will lead participants in procedures such as checking in (e.g. "How are you doing today?" before and after the circle) and breathing exercise.
  Interventions: Behavioral: Communal Drumming; Behavioral: Communal drumming recordings
- Drum Circle Control Group- Cohort 2 (Active Comparator): Control investigations will also be conducted to better understand the contribution communal drumming has on effects of anxiety and connectedness. All control investigations will take place in the same space and at the same frequency as the associated experimental arm but with no drumming. All participants will be asked to complete the same surveys and at the same frequency to those completed in the experimental arm.
  Interventions: Behavioral: Communal drumming recordings

INTERVENTIONS:
Behavioral: Communal Drumming — Communal drumming
  Arms: Drum Circle- Cohort 1
Behavioral: Communal drumming recordings — Recordings of drumming taken from the music made during a previous component of the study

SUMMARY:
Mental health vulnerability due to stress is increased America due to disproportionate effects of social factors such as racism, poverty, education, and criminal justice sentencing. Various meditation and mindfulness approaches have provided evidence of measured reductions in multiple negative dimensions of stress. However, the majority of these studies do not have an adequate representation of Persons of African Descent(PAD) or other marginalized groups and are not designed to be culturally relevant or community based. Music has been shown to alleviate multiple symptoms of stress and has been shown to be a preferred and effective support for meditation and mindfulness. However, its role in stress management in PADs engaged in meditation or mindfulness is seldom studied. This study aims to evaluate the effects of a community-based music mindfulness program on stress management in PAD community members with anxiety and depression during COVID19.

Component 2c. Drum Circle Study: Investigators will study the impact of participation in drum circles on anxiety and feelings of connectedness.

DETAILED DESCRIPTION:
The investigators also propose a study to investigate the effects of communal drumming in reducing anxiety and increasing connectedness within drum circle community. Investigators hypothesize that these intervention will lead to reductions in scores on stress scales and will provide preliminary data for studies evaluating these types of community programs as an adjunct to the standard of care.

Individuals who attend periodic (i.e. weekly) drum circles will be recruited to join an 8-week paradigm. Drum circle sessions may audio recorded and participants will be informed of this during the consent process. Participants may be asked to undergo Electroencepholography, functional Near Infrared Spectroscopy, and/or other physiological measures before, during, and after the circles. Upon completion of the experiments, participants will be asked to take part in a focus group that will provide valuable feedback on their experience with the mindfulness intervention. Focus groups will last 30-minutes to 1 hour and will occur in-person.

ELIGIBILITY:
Inclusion Criteria:

* ages 16 and older

Exclusion Criteria:

* ages 15 and younger

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Rating of Absorption in music pre vs post sessions | Baseline on day of study visit before drum circle, during drum circle (45min), 30 min after music listening
  These ratings are classified on a scale from 0 to 1, with 0 indicating no absorption and 1 indicating complete absorption.

SECONDARY OUTCOMES:
Altered States of Consciousness Rating Scale | Baseline on day of study visit before drum circle, during drum circle (45min), 30 min after music listening
  This scale has 94 statements and below each statement is a line with the endpoints "No, not more than usually" and "Yes, much more than usually." Each participant will rate to what extent the statements apply to their particular experience, compared to normal waking consciousness, by making a vertical mark on the line below the statements. Normal waking consciousness corresponds to a mark at the very left end of the scale, i.e.: "No, not more than usually."

CONTACTS AND LOCATIONS:
Overall Officials: AZA Allsop, MD, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - BLOOM, New Haven, Connecticut
  - Musical Intervention Studios, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
De-identified, aggregate data will be shared through pre-prints, publications, and community town hall meetings.